CLINICAL TRIAL: NCT00343954
Title: Phase 1 Pharmacokinetic and Pharmacodynamic Responses to Oral L-Citrulline in Patients With Sickle Cell Disease
Brief Title: PK and PD Responses to Oral L-Citrulline in Patients With Sickle Cell Disease
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Angiogenix (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ANGX-3227-01
Record Dates: First submitted 2006-06-21; First posted 2006-06-23 (Estimated); Last update posted 2006-06-23 (Estimated); Status verified 2006-06

CONDITIONS: Sickle Cell Disease
Keywords: sickle cell disease
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Citrulline

INTERVENTIONS:
Drug: L-citrulline tablets, 1000 mg

SUMMARY:
To evaluate PK and PD responses to L-citrulline given orally for four weeks to patients with sickle cell disease who are otherwise healthy.

DETAILED DESCRIPTION:
Phase 1, single center, open label, multiple-dose study consisting of a screening period followed by four weeks of treatment. At least 12 male and female patients, 10 years of age or older, with sickle cell disease but otherwise healthy, will be enrolled in the study.

PK measurements include plasma concentrations of L-citrulline, L-arginine, L-ornithine, and L-proline following the first dose of orally administered L-citrulline and after four weeks of twice daily administration of the drug.

PD measurements include intercellular and vascular adhesion molecules (ICAM, VCAM, and E-selectin), surrogate markers of sickle cell disease activity, and PAT, a measurement of vascular function.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 10 years of age or older on the day of dosing, and generally healthy as determined by medical history, physical examination, and laboratory test values
2. Diagnosis of sickle cell anemia (Hb SS)
3. For female of child-bearing potential, a negative serum pregnancy test and using an adequate method of contraception
4. Has signed and received a copy of the written informed consent form approved by the investigator's Institutional Review Board (IRB), understands the purposes and risks of the study and agrees to follow the restrictions and schedule of procedures as defined by this protocol

Exclusion Criteria:

1. History of sickle-cell-related pain crisis within two weeks of study
2. Pregnant or breast feeding
3. Transfusion within last 90 days
4. Creatinine >1.5 X upper limit of normal
5. SGPT > 2 X upper limit of normal
6. History of allergic reaction to arginine or citrulline product
7. Requires chronic medication other than study drug that cannot be discontinued during the study period
8. Unable to take or tolerate oral medications
9. Unreliable venous access
10. Noncompliant with regular care
11. Participation in an investigational drug or medical device study within previous 30 days
12. In the opinion of the investigator is not a good candidate for participation in the study

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12

PRIMARY OUTCOMES:
PK and PD responses to L-citrulline
Endpoints will be determined as change from baseline

SECONDARY OUTCOMES:
Assessment of safety and tolerability of L-citrulline,

CONTACTS AND LOCATIONS:
Overall Officials: Lakshmanam Krishnamurti, MD, Principal Investigator — Children's Hospital of Pittsburgh, Univ. of Pittsburgh Medical Center
Locations (1):
- Children's Hospital of Pittsburgh of the University of Pittsburgh Medical Center Health System, Pittsburgh, Pennsylvania, United States